CLINICAL TRIAL: NCT00218790
Title: The Effects of Hemodialysis on the Sleep/Wake Cycle
Brief Title: The Effects of Cool Dialysate on the Sleep/Wake Cycle in Patients on Chronic Hemodialysis - "The Sleep Cool Study"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Kathy P. Parker, PhD, RN, FAAN, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0602-2002a; R01NR004340 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2005-09

CONDITIONS: End-stage Renal Disease
Keywords: Sleep; Renal failure; Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): The control group received standard dialysis at a temperature of 37 degrees Celcius
- Experimental group (Experimental): Subjects in the experimental group received cool dialysate during treatment
  Interventions: Procedure: Cool Dialysate

INTERVENTIONS:
Procedure: Cool Dialysate — Decreased temperature of the dialysis bath
  Arms: Experimental group

SUMMARY:
A major component of this study is to test a novel application for a safe, non-pharmacologic, cost-effective intervention that is already in use in clinical practice - using cool dialysate during hemodialysis to help stabilize the sleep/wake cycle of chronic hemodialysis patients. We will also evaluate its effects on selected sleep-related physiologic, psychological, behavioral, and general health outcomes.

DETAILED DESCRIPTION:
Preliminary results demonstrate that, after one treatment, using cool dialysate instead of warm dialysate markedly normalized the rhythm of body temperature and improved indices on nocturnal sleep quantity and quality. Therefore, a major component of this study is to test a novel application for a safe, non-pharmacologic, cost-effective intervention that is alreay in use in clinical practice - using cool dialysate during hemodialysis to help stabilize the sleep/wake cycle of chronic hemodialysis patients. We will also evaluate its effects on selected sleep-related physiologic, psychological, behavioral, and general health outcomes.

To test the efficacy of this intervention, a randomized, single-blinded, pretest-posttest, control group design is being used. The major independent variable is dialysate temperature. The major dependent variables are measures of sleep, body temperature, rest/activity patterns, and general health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All races, cause of renal failure is diabetes, hypertension, glomerulonephritis, or polycystic kidney disease; ability to read and write in English; clinically stable.

Exclusion Criteria:

* Current use of sleeping medication; history of alcoholism or drug abuse; brain disease; severe hypertension; severe heart disease; low functional level

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
total sleep time | 9months
  amount of time slept per night

SECONDARY OUTCOMES:
quality of life | 9 months
  Quality of life as defined by the Ferrans and Powers QOL Inventory

OTHER OUTCOMES:
Comfort | 9 months
  Self-reported comfort as measured by a Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Kathy P. Parker, PhD,RN,FAAN, Principal Investigator — Emory University, Nell Hodgson Woodruff School of Nursing
Locations (2):
- United States (2):
  - Emory affiliated hemodialysis units, Atlanta, Georgia
  - Emory University affiliated hemodialysis units, Atlanta, Georgia

REFERENCES:
- [Background] Parker KP, Bliwise DL, Bailey JL, Rye DB. Polysomnographic measures of nocturnal sleep in patients on chronic, intermittent daytime haemodialysis vs those with chronic kidney disease. Nephrol Dial Transplant. 2005 Jul;20(7):1422-8. doi: 10.1093/ndt/gfh816. Epub 2005 Apr 19. PMID 15840682
- [Background] Lee KA, Landis C, Chasens ER, Dowling G, Merritt S, Parker KP, Redeker N, Richards KC, Rogers AE, Shaver JF, Umlauf MG, Weaver TE. Sleep and chronobiology: recommendations for nursing education. Nurs Outlook. 2004 May-Jun;52(3):126-33. doi: 10.1016/j.outlook.2003.12.002. No abstract available. PMID 15197361
- [Background] Parker KP, Kutner NG, Bliwise DL, Bailey JL, Rye DB. Nocturnal sleep, daytime sleepiness, and quality of life in stable patients on hemodialysis. Health Qual Life Outcomes. 2003 Nov 21;1:68. doi: 10.1186/1477-7525-1-68. PMID 14633280
- [Background] Parker KP. Sleep disturbances in dialysis patients. Sleep Med Rev. 2003 Apr;7(2):131-43. doi: 10.1053/smrv.2001.0240. PMID 12628214